CLINICAL TRIAL: NCT07208383
Title: Awareness, Knowledge and Behavioral Seeking of Gynaecological Problems
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chung Pui Wah Jacqueline, Associate Professor, Chinese University of Hong Kong
Other Study IDs: 2025.449
Record Dates: First submitted 2025-09-18; First posted 2025-10-06 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Gynecologic Disease
MeSH Terms: conditions — Genital Diseases, Female | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with gynecological problems: Gynecological patients aged between 13-60 years old, who have undergone or will seek medical service regarding their gynaecological problem, PCOS, endometriosis, miscarriage, or infertility, or attending gynecological clinics in the Prince of Wales Hospital.
  Interventions: Other: Questionnaire
- General public: For the General Public: Women aged 13-60 years old residing in Hong Kong, recruited through online platforms.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire to examine awareness, knowledge, and help-seeking behaviors among gynecological patients and the general public

SUMMARY:
This study seeks to fill this gap by examining awareness, knowledge, and help-seeking behaviors among gynecological patients and the general public. By comparing these groups, the study will identify disparities in knowledge and barriers to care, providing insights for targeted interventions to improve women's health outcomes in Hong Kong.

DETAILED DESCRIPTION:
In Hong Kong, limited health literacy and cultural taboos around discussing reproductive health may exacerbate these issues, particularly among younger women or those with lower socioeconomic status.

In Hong Kong, the interplay of Western and Chinese cultural values may create unique behavioral patterns, such as reliance on Traditional Chinese Medicine for gynecological issues or avoidance of medical care due to embarrassment. However, there is a lack of comprehensive data on how these factors specifically affect women with PCOS, endometriosis, miscarriage, or infertility in Hong Kong.

This study seeks to fill this gap by examining awareness, knowledge, and help-seeking behaviors among gynecological patients and the general public. By comparing these groups, the study will identify disparities in knowledge and barriers to care, providing insights for targeted interventions to improve women's health outcomes in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

Aged between 13 and 60 years old

Exclusion Criteria:

-Patients unable to provide consent/assent (i.e. significant psychiatric problems/cognitive delay)

Ages: 13 Years to 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: Gynecological patients aged between 13-60 years old, who have undergone or will seek medical service regarding their gynaecological problem, PCOS, endometriosis, miscarriage, or infertility, or attending gynecological clinics For the General Public: Women aged 13-60 years old residing in Hong Kong
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2035-08-31 (Estimated); Study Completion 2037-08-31 (Estimated)

PRIMARY OUTCOMES:
Awareness and knowledge about PCOS, endometriosis, miscarriage, and infertility | through study completion, an average of 1 year
  The level of awareness and knowledge about PCOS, endometriosis, miscarriage, and infertility among gynecological patients and the general public in Hong Kong will be assessed by the designated questionnaire.

SECONDARY OUTCOMES:
Behavioral patterns and barriers in seeking help for these gynecological problems | through study completion, an average of 1 year
  Their behavioral patterns and barriers in seeking help for these gynecological problems will be assessed by the designated questionnaire.
Awareness, knowledge, and help-seeking behaviors | through study completion, an average of 1 year
  Differences in awareness, knowledge, and help-seeking behaviors between gynecological patients and the general public will be assessed by the questionnaire.
Influence of socio-cultural and demographic factors | through study completion, an average of 1 year
  The influence of socio-cultural and demographic factors on awareness and help-seeking behaviors will be assessed by the designated questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Pui Wah Jacqueline Chung, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Obstetrics & Gynaecology The Chinese University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided